CLINICAL TRIAL: NCT03523767
Title: Effect of Systemic Inflammation on Emotion and Cognition in Patients With Mood Disorder - A Vaccine Study
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Early termination related to COVID pandemic
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Sudhakar Selvaraj, Sudhakar Selvaraj, MBBS., DPhil (Oxon)., MRCPsych, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: HSC-MS-16-0496
Record Dates: First submitted 2018-05-01; First posted 2018-05-14 (Actual); Last update posted 2023-04-04 (Actual); Status verified 2023-03

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Saline Solution

STUDY DESIGN:
Intervention Model Description: In this double blind crossover design, each participant will receive saline injection or typhoid vaccine injection at the first study visit, and will then receive the other injection at the second study visit.
Who Masked: Participant, Outcomes Assessor
Masking Description: The study clinician/ nurse will be aware of the nature of the injection. The study subjects and researcher collecting/analyzing the data will remain blinded to the intervention due to the possible confounding effects of the participant expectations and researcher analyzing the data.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Typhoid Vaccine, then Normal Saline (Experimental): 0.5 ml of S.typhi injection, then 0.5 ml of normal saline injection
  Interventions: Biological: S.typhi Injection; Biological: Normal Saline Injection
- Normal Saline, then Typhoid Vaccine (Placebo Comparator): 0.5 ml of normal saline injection, then 0.5 ml of S.typhi injection
  Interventions: Biological: S.typhi Injection; Biological: Normal Saline Injection

INTERVENTIONS:
Biological: S.typhi Injection — 0.5 ml of S.typhi injection
Biological: Normal Saline Injection — 0.5 ml of normal saline injection

SUMMARY:
The purpose of this pilot study is to investigate and compare the effect of a mild inflammatory stimulus (typhoid vaccine) on immune response, mood and cognition in healthy volunteers compared to patients with history Major Depressive Disorder (MDD) (not currently depressed and no symptoms of depression in the past 6 months).

DETAILED DESCRIPTION:
Study design: In this double blind randomized crossover design, each participant will receive saline injection or typhoid vaccine injection at the first study visit, and will then receive the other injection at the second study visit. All participants will undergo study procedures (clinical and imaging) in two separate sessions after each injection given at least 7 days apart (within 10-14 days).

Baseline blood samples will be taken and vital signs will be measured. Participants will be asked to complete the mood questionnaires and computerized reward tasks. Then, injections of normal saline will be administered intramuscularly in the deltoid muscle. At 1.5h, 3h, 4h and 6h after the injection, the subjects will complete the mood questionnaires and vital signs will be assessed. The computer based task will be repeated at 3h.

Between3h and 6h after the injection blood samples will be collected for cytokines measurement. At 4h, a structural magnetic resonance imaging (MRI), and Functional magnetic resonance imaging (fMRI) will be done.

Follow up visits/calls with the patients will be set to check their physical and mood status.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers, male or female; aged 18-65
* Subjects with history of Major depression (currently asymptomatic - symptom free for more than 6 months)
* Medication free, if not feasible being on antidepressants will be allowed

Exclusion Criteria:

* Volunteers who received this vaccine within 3 years or any other vaccine within 3 months
* Patients with existing inflammatory conditions (connective tissue disorder, autoimmune conditions, neoplastic disease, chronic infections, etc.)
* Patients with acute viral or bacterial infection
* Hospitalized patients
* Patients in acute phase of illness
* Current active medical condition that affect brain anatomy, neurochemistry, or function, e.g. liver insufficiency, kidney insufficiency, cardiovascular problems, systemic infections, cancer, hypothyroidism, auto-immune diseases, and any brain disorder (seizure disorder, stroke, dementia, degenerative neurologic diseases)
* History of any brain diseases, including seizures, stroke, meningitis, encephalitis, dementia, degenerative brain diseases, and serious head injury with loss of consciousness
* Family history of hereditary neurologic disorder
* Floating metallic objects in the body
* Pregnancy
* Exposure to regular use of anti-inflammatory drugs in the last one month
* Excessive exercise, consumption of caffeinated beverages or alcohol, high-fat meals 12 hours before testing
* History of tobacco, alcohol, or drug abuse or dependence.
* History of allergic reaction to vaccination or serious allergic reaction to shellfish or egg allergy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2018-02-07 (Actual); Primary Completion 2020-02-07 (Actual); Study Completion 2020-02-07 (Actual)

PRIMARY OUTCOMES:
Change in Inflammation as indicated by cytokines | baseline, 3-6 hours post-injection
  To compare proinflammatory cytokines (e.g. IL-6, TNF-α, etc) concentration between the experimental (receiving S.typhi vaccine) and the control group (receiving normal saline).
Change in depressed mood as indicated by Hamilton Depression Rating Scale (HAM-D) score | baseline, 3-6 hours post-injection
  To compare the severity of mood symptoms (as scored on the Hamilton Depression Rating Scale) between the experimental and the control group. A score of 0-7 is generally accepted to be within the normal range (or in clinical remission), while a score of 20 or higher indicates at least moderate severity of depressive symptoms. Scores range from 0-53.
Level of prefrontal, limbic and striatal cortex activation as indicated by fMRI | 3-6 hours post-injection
  Compare prefrontal cortex response to reward anticipation between the experimental and the control group, using fMRI

CONTACTS AND LOCATIONS:
Overall Officials: Sudhakar Selvaraj, 7134862627, Principal Investigator — Prinicpal Investigator
Locations (1):
- Sudhakar Selvaraj, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No